CLINICAL TRIAL: NCT00755040
Title: Randomized Placebo Controlled Double Blind Study of Restasis Versus Placebo in Primary Prevention of Ocular GVHD After Allogeneic Stem Cell Transplantation
Brief Title: Cyclosporine Eye Drops in Preventing Graft-Versus-Host Disease of the Eye in Patients Who Have Undergone Donor Stem Cell Transplant for Hematologic Cancer or Bone Marrow Failure Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Madan Jagasia, MD, Associate Professor of Medicine; Director, Outpatient Transplant Program; Section Chief, Hematology and Stem Cell Transplant; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VICC BMT 0766; P30CA068485 (NIH); VU-VICC-BMT-0766; VU-080786
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: graft versus host disease; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ocular Cyclosporine (Restasis) (Experimental): Patients receive cyclosporine ophthalmic emulsion (Restasis®) drops in each eye twice daily for up to 1 year after transplant.
  Interventions: Drug: cyclosporine ophthalmic emulsion
- Placebo (Placebo Comparator): Patients receive placebo ophthalmic drops in each eye twice daily for up to 1 year after transplant.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion — Given as eye drops
  Arms: Ocular Cyclosporine (Restasis)
Other: placebo — Given as eye drops
  Arms: Placebo

SUMMARY:
RATIONALE: Cyclosporine eye drops may prevent graft-versus-host disease of the eye in patients who have undergone donor stem cell transplant for hematologic cancer or bone marrow failure disorder.

PURPOSE: This randomized phase I trial is studying how well cyclosporine eye drops work in preventing graft-versus-host disease of the eye in patients who have undergone donor stem cell transplant for hematologic cancer or bone marrow failure disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy of cyclosporine ophthalmic emulsion (Restasis®) in the prevention of ocular graft-versus-host disease in patients who have undergone allogeneic stem cell transplantation for hematologic malignancies or bone marrow failure disorders.

Secondary

* To correlate the Ocular Surface Disease Index with clinical ophthalmologic examination.

OUTLINE: This is a multicenter study. Patients are stratified according to age, type of transplant (related vs unrelated), and intensity of transplant (ablative vs other). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclosporine ophthalmic emulsion (Restasis®) drops in each eye twice daily for up to 1 year after transplant.
* Arm II: Patients receive placebo ophthalmic drops in each eye twice daily for up to 1 year after transplant.

Patients in both arms may also receive artificial tear drops at least twice daily as clinically necessary.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 18 years at time of enrollment
* Day 80-120 after first allogeneic stem cell transplant for hematologic malignancies or -marrow failure disorder at time of study enrollment
* Signed informed consent
* Willing to adhere to protocol requirements

Exclusion criteria:

* history of non-compliance
* diagnosis of ocular GVHD at time of study enrollment
* documented dry eye prior to onset of stem cell transplant
* significant non- GVHD ocular problems that precludes participation in study
* life expectancy of lesser than 6 months at time of enrollment (viz. grade 4 acute GVHD, florid progression or relapse of underlying disease)
* history of documented ocular infections prior to stem cell transplant or during transplant (i.e. history of herpetic keratitis)
* females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Norwestern Memorial Hospital, Chicago, Illinois
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Dietrich-Ntoukas T, Cursiefen C, Westekemper H, Eberwein P, Reinhard T, Bertz H, Nepp J, Lawitschka A, Heiligenhaus A, Seitz B, Messmer EM, Meyer-ter-Vehn T, Basara N, Greinix H, Datiles MB, Lee SJ, Pavletic SZ, Wolff D. Diagnosis and treatment of ocular chronic graft-versus-host disease: report from the German-Austrian-Swiss Consensus Conference on Clinical Practice in chronic GVHD. Cornea. 2012 Mar;31(3):299-310. doi: 10.1097/ICO.0b013e318226bf97. PMID 22157574
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive cyclosporine ophthalmic emulsion (Restasis®) drops in each eye twice daily for up to 1 year after transplant.
  cyclosporine ophthalmic emulsion: Given as eye drops
- Arm II: Patients receive placebo ophthalmic drops in each eye twice daily for up to 1 year after transplant.
  placebo: Given as eye drops
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 83 | 81
Completed | 40 | 47
Not Completed | 43 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocular Cyclosporine (Restasis) | Placebo | Total
Number analyzed (Participants) | 83 | 81 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 75 | 156
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (12.458) | 49 (11.707) | 49 (12.062)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 73
  Male | 49 | 42 | 91
Region of Enrollment [Number; unit: participants]
  United States | 83 | 81 | 164

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Develop Ocular GVHD While on Study in the Two Arms (Ocular Cyclosporine (Restasis) vs. Placebo)
Description: Data analysis will be performed on an intention-to-treat basis. Logistic regression will be used to estimate the odds ratio and 95% confidence interval of the two treatment groups with the adjustment of baseline covariates. Outcome comparisons for categorical/dichotomous variables will be assessed by 2 test or Fisher's exact test where expected cell frequencies were <5; continuous variables will be compared by X/2 test or by Mann-Whitney U test where the data are strongly skewed.
Time Frame: Up to 2 years after transplantation
Population: Number of patients that develop ocular GVHD while on study
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 83 | 81
participants | 9 | 8
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p > 0.99, Fisher Exact; Odds Ratio (OR) = 1.11

2. Secondary Outcome: Numerical Score of Ocular Surface Disease Index (OSDI) and Development or Lack of Ocular GVHD (by Ophthalmologic Examination) as Measured by Odds Ratio in a Linear Regression Model.
Description: OSDI is a patient reported questionnaire consisting of 12 questions which are scored from 0 to 4. The total scored is computed and depending on the number of questions answered scores are computed which are then categorized into mild, moderate or severe dry eye symptoms. This tool should adequately reflect the morbidity of the dry eye symptoms.
Time Frame: 1 year after transplant
Population: Not collected/analysed due to staffing constraints
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 3/83 | 7/81
Other Adverse Events (participants affected / at risk) | 49/83 | 18/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=83) | Arm II (N=81)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 3 (3) | 4 (4) — Relapse of underlying disease
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Blood/Bone Marrow Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=83) | Arm II (N=81)
Burning (Eye disorders) | 31 (49) | 9 (18)
Red eye (Eye disorders) | 13 (13) | 18 (22)
Discharge (Eye disorders) | 9 (13) | 8 (8)
Excessive tearing (Eye disorders) | 14 (20) | 15 (21)
Eye pain (Eye disorders) | 5 (6) | 6 (6)
Foreign Body Sensation (Eye disorders) | 5 (5) | 8 (9)
Itching (Eye disorders) | 16 (20) | 9 (13)
Stinging (Eye disorders) | 17 (22) | 8 (9)
Visual disturbance (Eye disorders) | 13 (14) | 18 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No